CLINICAL TRIAL: NCT04850872
Title: PLAYwithHEART: Development and Feasibility Study of a Program for the Promotion of Acceptance and Cooperation Skills for Adolescent Athletes
Brief Title: PLAYwithHEART: PLAY With Happiness, Engagement, Acceptance, and Respect With Your Team
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Coimbra (Other)
Responsible Party: Principal Investigator, Sara Oliveira, MS, University of Coimbra
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: CINEICC; SFRH/BD/143410/2019 (Other Grant/Funding Number: Fundação para a Ciência e Tecnologia)
Record Dates: First submitted 2021-04-14; First posted 2021-04-20 (Actual); Last update posted 2024-03-21 (Actual); Status verified 2024-03

CONDITIONS: Adolescents; Athletes

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental (Experimental): PLAYwithHEART Programme is a manualized mindfulness, acceptance, and compassionate-based group intervention for adolescent competitive athletes. It included 8 weekly group sessions, 45 minutes each, run in small groups (ranging from 8 to 12 participants). Participants of this group complete also self-report measures.
  Interventions: Behavioral: PLAYwithHEART Programme for adolescent athletes
- Control (No Intervention): Participants of control group do not receive the intervention Programme (PLAYwithHEART), nor any other program, and only complete self-report measures.

INTERVENTIONS:
Behavioral: PLAYwithHEART Programme for adolescent athletes — PLAYwithHEART programme for adolescent athletes is an intervention programme based on Mindfulness, Acceptance, and Compassion for adolescent athletes
  Arms: Experimental

SUMMARY:
This investigation aims to apply and test the feasibility of a structured Program for young athletes. PLAYwithHEART is a program for promoting acceptance and cooperation skills in adolescent athletes. This group application program comprises eight weekly sessions and aims to decrease levels of sport anxiety, and increase the psychological quality of life of young athletes, by promoting skills inherent to an affiliation mentality (mindfulness, acceptance, and compassion), as an alternative to a social ranking mentality (based on maladaptive processes, such as shame and self-criticism), to deal with the challenges and demands of the sport context.

DETAILED DESCRIPTION:
The sample will include young athletes of different sports with ages ranged 12 to 18 years old. The principal investigator will recruit participants through contact with different sports clubs in Portugal. Athletes who demonstrate interest will go through a Screening interview (previously authorized by your legal guardian) by a licensed psychologist that aims explain the structure and arms of the investigation, to collect demographic data, and whether the athlete meets the inclusion criteria for the study. Athletes who meet the inclusion criteria and demonstrate interest in participating in the study, will sign an informed consent.

All ethical requirements for research with humans are guaranteed. Afterwards, participants will be allocated in two groups (experimental and control group). Additionally, the experimental group will enroll in the PLAYwithHEART programme, also provided by a licensed psychologist and a co-therapist.

Both groups will concurrently complete a protocol of self-report measures (to measure: a) psychological processes; b) quality of life and sports anxiety. These assessments will occur in three different times: before the start of the PLAYwithHEART programme (M0), after the final session of the programme (M1), and 6 months after that (M2).

ELIGIBILITY:
Inclusion Criteria:

* adolescent competitive athletes
* presentation of the informed consent signed by the participant and respetive legal guardian
* availability to participate in the 8 sessions of the PLAYwithHEART Programme
* inexistence of cognitive difficulties that interfere in completing self-response measures
* not being under psychological / psychiatric appointments

Exclusion Criteria:

* no presentation of the informed consent signed by the participant and respetive legal guardian
* unavailability to participate in the 8 sessions of the PLAYwithHEART Programme
* existence of cognitive difficulties that interfere in completing self-response measures
* being under psychological / psychiatric appointments

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 50 (Actual)
Dates: Start 2020-02-01 (Actual); Primary Completion 2024-08-01 (Estimated); Study Completion 2024-08-01 (Estimated)

PRIMARY OUTCOMES:
Changes in Quality of Life | From baseline to 6-months follow-up
  Measured by the The KIDSCREEN-10 quality of life measure for children and adolescents - higher levels mean a better outcome
Changes in competitive anxiety | From baseline to 6-months follow-up
  Measured by the Sport Anxiety Scale (SAS-2) - lower levels mean a better outcome

SECONDARY OUTCOMES:
Changes in Mindfulness | From baseline to 6-months follow-up
  Measured by the Children´s Acceptance and Mindfulness Measure (CAMM) - higher levels mean a better outcome
Changes in Psychological Inflexibility | From baseline to 6-months follow-up
  Measured by the Avoidance and Fusion Questionnaire for Youth (AFQ-Y) - lower levels mean a better outcome
Changes in Self-compassion | From baseline to 6-months follow-up
  Measured by the Self-Compassion Scale (SCS-A) - higher levels mean a better outcome
Changes in shame | From baseline to 6-months follow-up
  Measured by the External and Internal Shame Scale for adolescents (EISS-A). Lower scores mean a better outcome
Changes in self-criticism | From baseline to 6-months follow-up
  Measured by the Forms of self-criticizing/attacking and self-reassuring scale (FSCRS-A) - lower scores in self-criticising mean a better outcome

CONTACTS AND LOCATIONS:
Overall Officials: Sara Oliveira, MS, Principal Investigator — University of Coimbra
Locations (1):
- Different sports clubs in Portugal, Coimbra, Portugal